CLINICAL TRIAL: NCT05569668
Title: Neoadjuvant Chemotherapy Compared With Surgery for Esophageal Carcinoma: A Missing Evidence and A Retrospective Case-control Study
Brief Title: Neoadjuvant Chemotherapy Compared With Surgery for Esophageal Carcinoma
Status: Completed | Type: Observational
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: HCH2101
Record Dates: First submitted 2022-10-02; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Esophagus Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Paclitaxel; Platinum Compounds

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neoadjuvant chemotherapy group: Standard NAC comprised 2 cycles. Platinum plus paclitaxel or docetaxel was repeated once every 3 weeks. Cis-platinum was administered at a total dose of 75 mg/m2 by continuous infusion on d1 or equal divided on Days 2-4 or Days 1-3. Paclitaxel, 175 mg/m2, d1, or paclitaxel, 87.5 mg/m2, d1, d8. If the docetaxel was adopted, it was given as 75 mg/m2 on Day 1. Then surgery----esophagectomy and two-field extensive mediastinal lymphadenectomy. After surgery, there might be a adjuvant chemotherayp for pathologically positive lymph nodes patients.
- Primary surgery group: The patients would receive primary surgery----esophagectomy and two-field extensive mediastinal lymphadenectomy. After surgery, there might be a adjuvant chemotherayp for pathologically positive lymph nodes patients. .
  Interventions: Drug: Paclitaxel- and platinum-based chemotherapy

INTERVENTIONS:
Drug: Paclitaxel- and platinum-based chemotherapy — Neoadjuvant Chemotherapy
  Groups: Primary surgery group

SUMMARY:
Most ESCC received NAC in China without supportive evidence from local RCTs. The negative conclusion about NAC originated from Western countries in the 1990s. Whether two-field extensive mediastinal lymphadenectomy and paclitaxel/platinum-based chemotherapy results in better survival should be determined. As the highest ESCC incidence area worldwid, we tried to analyze this top with big data by using a single-center case-control retrospective PMS study. Paclitaxel- and platinum-based NAC combined with two-field of the extensive mediastinal lymphadenectomy might provide better survival benefits than primary esophagectomy for stage II/III SCC.

DETAILED DESCRIPTION:
Treatment Neoadjuvant Chemotherapy Standard NAC comprised 2 cycles. Platinum plus paclitaxel or docetaxel was repeated once every 3 weeks. Cis-platinum was administered at a total dose of 75 mg/m2 by continuous infusion on d1 or equal divided on Days 2-4 or Days 1-3. Paclitaxel, 175 mg/m2, d1, or paclitaxel, 87.5 mg/m2, d1, d8. If the docetaxel was adopted, it was given as 75 mg/m2 on Day 1.

Surgical Procedure At approximately 6-8 weeks after NAC, open (McKeown, left thoracic incision left cervical anastomosis) or MIE via thoracoscopy and/or laparoscopy was performed in the patients. Bilateral laryngeal recurrent nerve lymph node dissection was requested for every patient.

Comparisons between the NAC and primary surgery groups were performed using the chi-square test, Mann-Whitney U test and Fisher's exact test for categorical parameters after PMS. Kaplan-Meier curves and a Cox proportional hazards regression model were adopted to perform OS analysis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Esophageal Squamous Cell Carcinoma(ESCC) at Henan Cancer Hospital between January 1, 2015, and December 31, 2018 and the data was prospectively collected in the hubble of the LinkDoc data company
* Surgery performed in the thoracic surgery department
* No previous cancer treatment

Exclusion Criteria:

* Patients with secondary cancer were excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinical diagnosis of Esophageal Squamous Cell Carcinoma(ESCC) at Henan Cancer Hospital between January 1, 2015, and December 31, 2018
Sampling Method: Non-Probability Sample
Enrollment: 826 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
OS(overall survival) | From date of patient admission to the inpatient thoracic surgery department until the date of first documented death from any cause, assessed up to 100 months
  OS was defined as the first date of patient admission to the inpatient thoracic surgery department to the date of death from any cause.

SECONDARY OUTCOMES:
DFS(disease-free survival) | From date of patient admission to the inpatient thoracic surgery department until the date of first documented progression, assessed up to 100 months
  DFS was defined as the first day of patients admission to the inpatient department to the date of tumor recurrence confirmed by the follow-up tests.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zheng, PhD, MD, Principal Investigator — Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university
Locations (1):
- Henan Cancer Hospital (The Affiliated Cancer Hospital of Zhengzhou University), Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No